CLINICAL TRIAL: NCT00523393
Title: Prospective Influence of Bedtime Insulin Glargine on Mobilization and Function of Endothelial Progenitor Cells in Patients With Type 2 Diabetes: a Partially Double-Blind, Randomized, Three-Arm Unicenter Study
Brief Title: Prospective Influence of Bedtime Insulin Glargine on Mobilization and Function of Endothelial Progenitor Cells
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Dr. Per M. Humpert, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006-006573-24
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention)
- 2 (Experimental)
  Interventions: Drug: Insulin Glargin
- 3 (Active Comparator)
  Interventions: Drug: Human Insulin

INTERVENTIONS:
Drug: Insulin Glargin — Titration of bedtime insulin glargin aiming at normal morning fasting glucose
  Other Names: Lantus®, HOE901 (internal code number Sanofi-Aventis)
  Arms: 2
Drug: Human Insulin — Titration of bedtime human insulin aiming at normal morning fasting glucose
  Other Names: Insuman Basal®, HR1799(internal code number Sanofi-Aventis)
  Arms: 3

SUMMARY:
In this trial, it will be studied whether early addition of the long acting insulin analogue Glargine is capable of increasing the number and differentiation of endothelial progenitor cells (EPC) in patients with type 2 diabetes, which can be seen as a marker of vascular regenerative potential and cardiovascular risk. In addition, the effect of Glargine on microvascular function will be studied. This will be done using laser Doppler measurements of the skin; in addition, MRI of the heart will be performed which is capable of quantifying the perfusion reserve of the myocardium and additional functional aspects of ventricular function. A beneficial effect of early addition of bedtime Glargine on EPC and vascular as well as myocardial function in this study might argue for a change in the therapeutic approach in type 2 diabetes and possibly improve the cardiovascular outcome in patients affected.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Oral antidiabetic therapy
* Age 35 - 70
* 6,5%< HbA1c ≤ 9%
* Ability of subject to understand character and individual consequences of clinical trial
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception (Pearl Index < 1%, e.g. birth control pill) and negative blood pregnancy test
* 6,5%< HbA1c ≤ 9%
* Ability of subject to understand character and individual consequences of clinical trial
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception (Pearl Index < 1%, e.g. birth control pill) and negative blood pregnancy test

Exclusion Criteria:

* MODY
* Malignant disease
* Hematopoietic disorders
* Impairment of renal function (Serum creatinine > 1,5mg/dl)
* autoimmune disease
* treatment with immunosuppressive drugs
* Psychiatric disease
* Myocardial ischemia during previous 6 month
* Acute coronary syndrome
* pAVK IIb, III, IV (Fontaine-Ratschow)
* Erythropoietin treatment
* Glitazone treatment during two weeks before inclusion
* Insulin treatment during two weeks before inclusion
* Pregnancy and lactation
* History of hypersensitivity to the investigational product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational product
* Participation in other clinical trials and observation period of competing trials, respectively
* No subject will be allowed to enroll in this trial more than once.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Change of number of circulating EPC 4 weeks after start of therapy compared to baseline as detected by FACS analysis | 4 weaks of treatment

SECONDARY OUTCOMES:
Change of number of circulating EPC 4 as detected by in vitro outgrowth | 4 weeks, 4 months
Skin microvascular function (as measured by laser Doppler perfusion upon heat stimulation) | 4 months
Myocardial function and myocardial perfusion reserve as measured by MRI | 4 months
Intima-Media-Thickness | 4 months
Long-term Glucose control (HbA1c) | 4 weeks, 4 months
Short-term Glucose control (fasting glucose) | 4 weeks, 4 months
Markers of inflammation and vascular risk in diabetes | 4 weeks, 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Per M Humpert, Dr., Principal Investigator — University of Heidelberg, Dept. Medicine 1, Germany
Locations (1):
- University Clinics Heidelberg, Dept. Medicine1, Heidelberg, Germany

REFERENCES:
- [Derived] Oikonomou D, Kopf S, von Bauer R, Djuric Z, Cebola R, Sander A, Englert S, Vittas S, Hidmark A, Morcos M, Korosoglou G, Nawroth PP, Humpert PM. Influence of insulin and glargine on outgrowth and number of circulating endothelial progenitor cells in type 2 diabetes patients: a partially double-blind, randomized, three-arm unicenter study. Cardiovasc Diabetol. 2014 Oct 11;13:137. doi: 10.1186/s12933-014-0137-4. PMID 25300286